CLINICAL TRIAL: NCT03547128
Title: Iowa Fluoride Study/Iowa Bone Development Study
Acronym: (IFS/IBDS)
Status: Completed | Type: Observational
Sponsor: Steven M Levy (Other)
Responsible Party: Sponsor-Investigator, Steven M Levy, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 199112665
Record Dates: First submitted 2018-01-11; First posted 2018-06-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries; Dental Fluoroses; Bone Density
Keywords: fluoride; genetics; physical activity; diet
MeSH Terms: conditions — Dental Caries; Fluorosis, Dental; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary samples collected for DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parents with newborns recruited from 1992-5: Parents of newborns recruited from 8 Iowa hospitals in 1992-5

SUMMARY:
A cohort of newborns was recruited for the Iowa Fluoride Study from 1992-95 to assess the complex relationships among fluoride intakes, fluoride exposures, dental fluorosis, and dental caries. Detailed questionnaires were sent every 1.5-6 months concerning water sources, fluoride exposures, dietary intakes, etc. Standardized dental exams were conducted at ~ages 5, 9, 13, 17, and 23. At about age 5, participants were invited to join the offshoot Iowa Bone Development Study. Bone densitometry assessments were conducted at ages 5, 8, 11, 13, 15, 17, 19, and 23. These included Dual-energy X-ray Absorptiometry (DXA) of hip, lumbar spine, and whole body from age 5; peripheral Quantitative Computed Tomography (pQCT) of the radius and tibia from age 11; and Multi-Detector Computed Tomography (MDCT) of the tibia from age 19. Physical activity and other factors also were assessed longitudinally.

DETAILED DESCRIPTION:
A cohort of newborns was recruited for the Iowa Fluoride Study from 1992-95 to assess the complex relationships among fluoride intakes, fluoride exposures, dental fluorosis, and dental caries. Detailed questionnaires were sent every 1.5-6 months concerning water sources, fluoride exposures, dietary intakes, etc. Standardized dental exams were conducted at ~ages 5, 9, 13, 17, and 23. At about age 5, participants were invited to join the offshoot Iowa Bone Development Study. Bone densitometry assessments were conducted at ages 5, 8, 11, 13, 15, 17, 19, and 23. These included Dual-energy X-ray Absorptiometry (DXA) of hip, lumbar spine, and whole body from age 5; peripheral Quantitative Computed Tomography (pQCT) of the radius and tibia from age 11; and Multi-Detector Computed Tomography (MDCT) of the tibia from age 19. Physical activity and other factors also were assessed longitudinally.

ELIGIBILITY:
Inclusion Criteria:

* healthy newborn

Exclusion Criteria:

* not health newborn

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: newborns recruited from 8 Iowa hospitals postpartum
Sampling Method: Non-Probability Sample
Enrollment: 1882 (Actual)
Dates: Start 1992-03-01 (Actual); Primary Completion 1996-03-01 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
dental fluorosis-5 | age 5
  dental fluorosis exam results
dental fluorosis-9 | age 9
  dental fluorosis exam results
dental fluorosis-13 | age 13
  dental fluorosis exam results
dental fluorosis-17 | age 17
  dental fluorosis exam results
dental fluorosis-23 | age 23
  dental fluorosis exam results
dental caries-5 | age 5
  dental caries exam results
dental caries-9 | age 5
  dental caries exam results
dental caries-13 | age 9
  dental caries exam results
dental caries-17 | age 17
  dental caries exam results
dental caries-23 | age 23
  dental caries exam results
bone densitometry-5 | age 5
  DXA scans
bone densitometry-8 | age 8
  DXA scans
bone densitometry-11 | age 11
  DXA and pQCT scans
bone densitometry-13 | age 13
  DXA and pQCT scans
bone densitometry-15 | age 15
  DXA and pQCT scans
bone densitometry-17 | age 17
  DXA and pQCT scans
bone densitometry-19 | age 19
  DXA, pQCT, and MDCT scans
bone densitometry-23 | age 23
  DXA, pQCT, and MDCT scans

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Levy, dds, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: Yes
some data are available in NIH repository under DBGap
Time Frame: some past data are there now
  caries outcomes and explanatory factors
Access Criteria: contact PI for discussions and permissions

REFERENCES:
- [Derived] Marshall TA, Curtis AM, Cavanaugh JE, Warren JJ, Levy SM. Beverage Intakes and Toothbrushing During Childhood Are Associated With Caries at Age 17 Years. J Acad Nutr Diet. 2021 Feb;121(2):253-260. doi: 10.1016/j.jand.2020.08.087. Epub 2020 Oct 24. PMID 33109505
- [Derived] Marshall TA, Curtis AM, Cavanaugh JE, Warren JJ, Levy SM. Child and Adolescent Sugar-Sweetened Beverage Intakes Are Longitudinally Associated with Higher Body Mass Index z Scores in a Birth Cohort Followed 17 Years. J Acad Nutr Diet. 2019 Mar;119(3):425-434. doi: 10.1016/j.jand.2018.11.003. Epub 2019 Jan 9. PMID 30638821